CLINICAL TRIAL: NCT02674373
Title: Prognostic and Predictive Impact of Circulating Tumor DNA in Advanced and Localized Gastric Cancer Treatment
Brief Title: Prognostic and Predictive Impact of Circulating Tumor DNA in Gastric Cancer Treatment
Acronym: PLAGAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Association des Gastroentérologues Oncologues (Other)
Responsible Party: Principal Investigator, Dr. Aziz Zaanan, MD, PhD, Association des Gastroentérologues Oncologues
Other Study IDs: NI-GC-DNAc
Record Dates: First submitted 2015-12-08; First posted 2016-02-04 (Estimated); Last update posted 2016-02-04 (Estimated); Status verified 2016-02

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; biomarker; Circulating tumor DNA; Chemotherapy; Prognosis; Predictive
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — circulating tumor DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Localized gastric cancer: resectable tumor receiving a curative intent treatment.
- advanced gastric cancer: unresectable tumor treated with palliative chemotherapy

SUMMARY:
The evaluation of the chemotherapy efficacy for gastric cancer patients is usually evaluated by computer tomography scans with RECIST criteria that are performed every two months during the treatment. The management of treatment for gastric cancer needs the development of early biomarkers to evaluate the efficacy in order to avoid unnecessary toxicity in case of early chemotherapy resistance. In this prospective study, we will compare the monitoring of circulating tumor DNA with the results of CT scan according the RECIST criteria and the blood level of CEA and CA 19-9 tumor markers.

Thus, the objective of this study is to identify a prognostic and/or predictive biomarker of tumor response according to the tumor DNA circulating assessment in gastric cancer treatment, in order (i) to avoid an unnecessary toxicity of an ineffective treatment that it would be continued uselessly, (ii) and to allow a early changing to an alternative chemotherapy regimen.

DETAILED DESCRIPTION:
Introduction The cell lysis phenomena tumor releases DNA that can be detected in the blood and in other biological fluids such as lymph, urine or stool. An increase in plasma levels of tumor DNA is described in patients with cancer, and recently, monitoring of circulating tumor DNA that has been proposed as a relevant potential marker to assess the prognosis and the early response to treatment of colon or breast cancers (Dawson et al, 2013; Spindler et al, 2013; Tie et al, 2015). However, there is no data on the prognostic and predictive impact of circulating tumor DNA in context of gastric cancer treatment.

The aim of this study is to evaluate the correlation between the level of circulating tumor DNA and prognosis or response to treatment of localized and advanced gastric cancer.

Patients and Methods:

Three university hospitals of "Assistance Publique Hôpitaux de Paris" (AP-HP) will participate in this prospective study: European Georges Pompidou hospital, Pitié-Salpêtrière hospital and Cochin hospital. Inclusion criteria were all patients aged over 18 years with localized or advanced adenocarcinoma of gastric or gastro-oesophageal junction, histologically proven. The patients will be enrolled over a period of 2 years after receiving and signed a specific consent information form.

This is a non-interventional study who does not change the management of patients. There will be no additional invasive procedures to those already scheduled for routine care. Blood samples will be made at the time of chemotherapy sessions from the Huber needle previously implanted in the port-a-cath for the administration of chemotherapy agents.

The circulating tumor DNA is analyzed and quantified by sequencing proton from somatic genetic alterations identified in the tumor (Inserm Unit 775 UMR_S, Professor Pierre Laurent-Puig).

The data related to the patient (age at diagnosis, sex, weight, height, WHO performance status), tumor (tumor markers CEA and CA 19-9, date of diagnosis of gastric cancer, histological type and tumor differentiation, tumor stage, and metastatic sites) and treatment (resection of the primary tumor, date of surgery, chemotherapy protocol) will be collected anonymously. Monitoring data concern the efficacy of chemotherapy (tumor response, the date of disease progression, survival), as well as the possible dates of tumor recurrence or death.

The Statistical analysis will be based on a survival model in order to predict the responder or non-responder status, including parameters normally associated with risk of recurrence and death. The association between changing in circulating tumor DNA levels in responders and non-responders will be performed with a Cox model; the DNA circulating levels will be considered as a variable dependent of time. An estimation of 100 patients is planned for each cohort (localized and advanced diseases) with a recruitment period of approximately 2 years.

Expected Results

* For the cohort of patients with a localized tumor: loss (or decrease) in circulating tumor DNA after curative treatment for patients who do not exhibit tumor recurrence; OR no loss (or increase) in circulating tumor DNA after curative treatment in patients with tumor recurrence.
* For the cohort of patients with advanced tumor: early and significant increase in the level of circulating tumor DNA in non-responders to chemotherapy; OR early and significant reduction in the level of circulating tumor DNA in patients who respond to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients aged over 18 years
* histologically proven adenocarcinoma of gastric or gastro-oesophageal junction
* And receiving treatment:

  * For localized tumor stage: surgical resection associated with perioperative chemotherapy, adjuvant chemotherapy or adjuvant chemoradiotherapy
  * For advanced tumor stage: first-line palliative chemotherapy

Exclusion Criteria:

* All patients unable to undergo medical monitoring study for geographical, social or psychic reasons ;
* Patients under guardianship or unable to read, understand and sign the information sheet and consent form;
* Non-affiliated to the French social security institution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated for a histologically proven, localized or advanced adenocarcinoma of gastric or gastro-oesophageal junction, will be enrolled in this prospective cohort study after receiving and signed a specific consent information form.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Time from the start of treatment until progression disease (advanced tumor cohort) assessed up to 9 months, or recurrence (localized tumor) assessed up to 24 months
  PFS will be evaluated according to the circulating tumor DNA

SECONDARY OUTCOMES:
Tumor response rate | Tumor response rate according to the RECIST 1.1 criteria. This outcome measure will be assessed through study completion, an average of 6 months
  Tumor response rate will be evaluated according to the circulating tumor DNA
Overall survival (OS) | Time from the start of treatment until death assessed up to 24 months (advanced tumor cohort)
  OS will be evaluated according to the circulating tumor DNA

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Zaanan, MD, PhD, Principal Investigator — European Georges Pompidou Hospital, Paris, France
Locations (1):
- European Georges Pompidou Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No